CLINICAL TRIAL: NCT06750536
Title: Evaluating the Safety and Performance of the MiniLung Petite Kit in Neonatal and Pediatric Patients With Acute Respiratory and Cardiac Failure
Acronym: PETIT
Status: Recruiting | Type: Observational
Sponsor: Xenios AG (Industry)
Collaborators: Alcedis GmbH (Industry)
Responsible Party: Sponsor
Organization: Fresenius Medical Care Deutschland GmbH (Industry)
Other Study IDs: PMCF-MLP-01-EU
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Neonatal Aspiration Pneumonia; Acute Respiratory Failure; Acute Lung Injury
Keywords: Extracorporeal Membrane Oxygenation; Neonatal and pediatric patients; MiniLung petite kit
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MiniLung petite kit combined with the Xenios console — Veno-venous (VV) and veno-arterial (VA) Extracorporeal Membrane Oxygenation (ECMO) treatment will be performed using the MiniLung petite kit combined with the Xenios console according to their intended use and local standards/requirements.

SUMMARY:
This prospective observational study will evaluate the safety and performance of the MiniLung petite kit in neonatal and pediatric patients with acute respiratory and cardiac failure.

The main question it aims to answer is (study hypotheses):

Veno-venous (VV) and veno-arterial (VA) Extracorporeal Membrane Oxygenation (ECMO) using the MiniLung petite kit is safe and improves gas exchange (oxygenation and CO2 removal) and hemodynamic stabilization in neonatal and pediatric patients with severe acute respiratory and/or cardiopulmonary failure within 24 hours compared to the treatment before VV or VA ECMO initiation and maintain a life-sustaining condition.

ELIGIBILITY:
Inclusion criteria

* Informed consent signed and dated by parents or legal representative and investigator/authorized physician
* Patients ≥2- ≤8 kg bodyweight to be treated with the MiniLung petite kit
* Acute severe respiratory and/or cardiopulmonary failure with an ECMO indication

Exclusion criteria:

* Participation in an interventional clinical study during the preceding 30 days that could interfere with the ECLS therapy
* Previous participation in the same study
* Prematurity (<34 weeks gestational age)
* Hypersensitivity to heparin or known history of heparin induced thrombocytopenia (HIT)
* Impossibility of systemic anticoagulation

Max Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal and/or pediatric patients with severe acute respiratory and/or cardiopulmonary failure treated with VV or VA ECMO.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Oxygenation Index | Baseline and during the intervention every 24 hours until a maximum of 29 days
  Longitudinal assessments of continuous outcomes will be analyzed by treatment day using mixed models for repeated measures (MMRM), with ECMO mode as a fixed factor (except for analyses performed within the subsets defined by ECMO mode) and the baseline value of the primary endpoint (Oxygenation Index) as a covariate.
  Within-subject differences between baseline and subsequent visits will be tested using contrasts. The comparison between baseline and the first day on ECMO (initial effect) is considered as the primary outcome.

SECONDARY OUTCOMES:
Hemodynamic stabilization | Baseline and during the intervention every 24 hours until a maximum of 29 days
  Longitudinal assessments of continuous outcomes will be analyzed by treatment day using mixed models for repeated measures (MMRM), with ECMO mode as a fixed factor (except for analyses performed within the subsets defined by ECMO mode) and the baseline value of the secondary endpoint (Hemodynamic stabilization) as a covariate.
  Within-subject differences between baseline and subsequent visits will be tested using contrasts. The comparison between baseline and the first day on ECMO (initial effect) is considered as the secondary outcome of Hemodynamic stabilization.
Facilitate lung-protective ventilation in patients additionally receiving invasive mechanical ventilation | Baseline and during the intervention every 24 hours until a maximum of 29 days
  Longitudinal assessments of continuous outcomes will be analyzed by treatment day using mixed models for repeated measures (MMRM), with ECMO mode as a fixed factor (except for analyses performed within the subsets defined by ECMO mode) and the baseline value of the secondary endpoint (Lung-protective ventilation) as a covariate.
  Within-subject differences between baseline and subsequent visits will be tested using contrasts. The comparison between baseline and the first day on ECMO (initial effect) is considered as the secondary outcome of lung-protective ventilation.
Assessment of the frequency of complications | Baseline and during the intervention every 24 hours until a maximum of 29 days
  Longitudinal assessments of continuous outcomes will be analyzed by treatment day using mixed models for repeated measures (MMRM), with ECMO mode as a fixed factor (except for analyses performed within the subsets defined by ECMO mode) and the baseline value of the secondary endpoint (Frequency of complications) as a covariate.
  Within-subject differences between baseline and subsequent visits will be tested using contrasts. The comparison between baseline and the first day on ECMO (initial effect) is considered as the secondary outcome of frequency of complications.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Müller, Prof. Dr., Principal Investigator — University Hospital, Bonn
Locations (2):
- Germany (2):
  - Universitätsklinkum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Mannheim, Mannheim

IPD SHARING:
Plan to Share IPD: Undecided